CLINICAL TRIAL: NCT05296109
Title: Application of 3D Magnetic Resonance Neurogram Sequences for Evaluation of Intraparotid Facial Nerves in Patients With Parotid Neoplasm
Brief Title: Application of 3D MR Neurogram for Intraparotid Facial Nerves Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Leung Ho Sang, Resident and Honorary Clinical Tutor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CREC 2021.639
Record Dates: First submitted 2022-02-25; First posted 2022-03-25 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Parotid Neoplasms
MeSH Terms: conditions — Parotid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging group (Experimental): patients with parotid tumour being imaged
  Interventions: Diagnostic Test: Magnetic Resonance Imaging on 3T scanner (Magnetom Prisma, SIemens) with dedicated neurogram sequences (Constructive interference in steady state - CISS; Dual Echo Steady State - DESS)

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging on 3T scanner (Magnetom Prisma, SIemens) with dedicated neurogram sequences (Constructive interference in steady state - CISS; Dual Echo Steady State - DESS) — The MRI examination will consist of both conventional sequences for diagnosis of salivary gland neoplasms (including DWI and DCE-MRI), together with additional neurogram sequences. (please refer to attached protocol for list of sequences)

SUMMARY:
Parotid neoplasm consists of a wide range of benign and malignant lesions, and parotidectomy has been the mainstay for management of these neoplasms. Within the parotid gland there are branches of the intra-parotid facial nerves, which are tiny in calibre and are prone to injury to injury during operation. It has been reported in recent retrospective view that the incidence of temporary and permanent facial nerve injury were 9.2% and 5.2% respectively, the risk of which increased with old age, malignant tumour and revision surgery. Traditional the incidental of facial nerve injury is reduced by intra-operative facial nerve monitoring and surgical magnification, while imaging has limited role in aiding this purpose. However with advancement in MRI technique high resolution three-dimensional sequences (i.e. neurogram sequences) are available for better visualization of branches of facial nerves. The investigators would therefore aim to demonstrate additional efficacy of these techniques and also to compare with conventional 3D post-contrast anatomical imaging studies in the localization and visualization of the facial nerve branches in patients with tumour. With better pre-operative imaging, the investigators hope to reduce the chance of facial nerve injury in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with parotid tumour diagnosed on other imaging modalities (such as ultrasonography or computed tomography), with or without cytological diagnosis from fine needle aspiration, will be recruited from the ear, nose and throat specialty clinic.

Exclusion Criteria:

* Patients who are contraindicated to magnetic resonance imaging (such as due to underlying MRI incompatible metallic implants)
* Patient who are contraindicated to MRI contrast agents (such as advanced renal failure or previous severe allergic reaction)
* Patients who cannot cooperate for MRI scanning.
* Patients show are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
visualization of the major branches of the facial nerve on MRI sequences | At MRI scan before therapeutic intervention (operation or radiofrequency ablation)
  The degree which facial nerve and branches will be visualized, by a three-point scale to each facial nerve branch, after review by radiologist.
  Total score of facial nerve visualization will be calculated, per MRI sequence per patient.

SECONDARY OUTCOMES:
Diagnostic value of multi-parametric MRI | At MRI scan before therapeutic intervention (operation or radiofrequency ablation)
  The sensitivity, specificity and accuracy of MRI on distinguishing benign and malignant parotid tumours using DWI and DCE-MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Sang Leung, MBBS (HK), Principal Investigator — Department of Imaging and Interventional Radiology, Prince of Wales Hospital; Chiu Wing WInnie Chu, MD, FHKCR, Study Director — Department of Imaging and Interventional Radiology, Prince of Wales Hospital
Locations (1):
- Gerald Choa MRI Center, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared includes individual participant data that underlie the results reported in this article, after deidentification.
Supporting Information: Study Protocol
Time Frame: Within 3 years after publication of article.
Access Criteria: Proposals should be directed to lhs655@ha.org.hk. To gain access, data requestors will need to sign a data access agreement. Data are available for 3 years at CUHK research data repository. (https://researchdata.cuhk.edu.hk//)

DOCUMENTS (2):
  • Study Protocol (2022-06-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT05296109/Prot_002.pdf
  • Informed Consent Form (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT05296109/ICF_003.pdf